CLINICAL TRIAL: NCT03775083
Title: What Happens in Vegas: Identifying Opportunities to Expand an HIV Prevention Network to Improve PEP and PrEP Delivery
Brief Title: What Happens in Vegas: PEP to PrEP Opportunities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huntridge Family Clinic (Other)
Responsible Party: Principal Investigator, John Phoenix, Clinical Director, Huntridge Family Clinic
Other Study IDs: HFC018001
Record Dates: First submitted 2018-09-06; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Exposure to Human Immunodeficiency Virus (Event)
Keywords: PEP; nPEP; Post Exposure Prophylaxis; non occupational exposure to HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Currently approved medications — subjects will be treated according to current Department of Health and Human Services (DHHS) Center for Disease control and prevention (CDC), Society for Healthcare Epidemiology of American (SHEA guidelines for nPEP

SUMMARY:
Observational study looking at barriers to care for individuals seeking care, Post Exposure Prophylaxis (PEP) after an actual or perceived exposure to HIV. Following PEP treatment subjects will be asked about there intent to transition to Pre-Exposure Prophylaxis (PrEP) and surveyed about barriers to care or perceptions of care

DETAILED DESCRIPTION:
The primary objective of this study is to assess the rate of engagement in a PEP to PrEP HIV provider network for those patients presenting following a non-occupational HIV exposure.

The development of a referral network and intensive clinical follow up of PEP patients will result in more patients appropriately initiating PEP, being referred to appropriate follow up, and post exposure transition and maintaining on PrEP (if indicated) at completion of the PEP medications.

ELIGIBILITY:
Inclusion Criteria:

* Actual or perceived non-occupational exposure to HIV, by self report, within 72 hours of enrollment and referred for care
* able and willing to provide informed consent
* available for 12 months of post expoure follow-up Southern Nevada Ryan White defined service area

Exclusion Criteria:

* HIV+ at time of screeing via 4th genderation (Antibody/Antigen) testing
* Current PEP and/or PrEP product condrainidications as listed in the medication product insert.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV negative Men, Women, Transgender Men, Transgender Women age who self identify as having had an actual or perceived non-occupational exposure to HIV
  HIV negative Men, Women, Transgender Men, Transgender Women age who self identify at risk of acquisition of HIV after having had an actual or perceived non-occupational exposure to HIV
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
rate of engagement | from enrollment to day 90
  Assess the rate of engagement in a PEP to PrEP HIV prevention provider network for those patients presenting following a non-occupational HIV exposure

SECONDARY OUTCOMES:
characteristics | from enrollment through end of study for all participants
  Describe the characteristics of patients successfully engaging in HIV prevention via a patient collected survey using a qualtric survey.
barriers | from enrollment through end of study for all participants
  Identify and assess barriers to access to HIV prevention care including PEP in the period immediately following HIV exposure from a patient collected survey using a qualtric survey tool
Network characteristics | from enrollment through end of study for all participants
  Analyze the network characteristics that faciliate engagement in HIV prevention services from a patient collected survey using a qualtric survey tool
transition barriers | from enrollment through end of study for all participants
  Determine and assess to transitioning from PEP to PrEP from a patient collected survey using a qualtric survey tool
Retention | from enrollment through end of study for all participants
  Compare and contrast the barriers to access and ongoing retention to PrEP from a patient collected survey using a qualtric survey tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntridge Family Clinic, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No